CLINICAL TRIAL: NCT00585377
Title: AVF4236s: Bevacizumab (Avastin®) + Erlotinib as First-line Therapy for Stage IIIB/IV or Recurrent, Non-squamous Cell Lung Cancer
Brief Title: Bevacizumab (Avastin®) + Erlotinib as First-line Therapy for Stage IIIB/IV or Recurrent, Non-squamous Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI24377; AVF4236s:
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Bevacizumab and Erlotinib

INTERVENTIONS:
Drug: Bevacizumab and Erlotinib — Erlotinib 150 mg/day orally plus bevacizumab 15 mg/kg intravenously every 21 days
  Other Names: Bevacizumab: Avastin®; Erlotinib: Tarceva®

SUMMARY:
In an attempt to improve the therapeutic index for initial therapy of metastatic NSCLC, the combination of bevacizumab and erlotinib is being proposed as first-line treatment in place of conventional chemotherapy. This trial is intended to provide pilot data for a future randomized trial of this combination of targeted agents versus conventional chemotherapy for advanced NSCLC.

DETAILED DESCRIPTION:
The combination of Bevacizumab and Erlotinib show encouraging activity for patients with previously treated, non-small-cell lung cancer. In a phase I/II study of erlotinib and bevacizumab in patients with nonsquamous stage IIIB/IV NSCLC with one or more prior chemotherapy exposures, a recommended phase II dose was established at erlotinib 150 mg/day orally plus bevacizumab 15 mg/kg intravenously every 21 days (13) Forty patients were treated at the recommended Phase II dose. The median age was 59 years (range, 36 to 72 years), 21 were female, 30 had adenocarcinoma histology, nine were never-smokers, and 22 had > or = two prior regimens (three patients had > or = four prior regimens). The most common adverse events were mild to moderate rash, diarrhea, and proteinuria. No pharmacokinetic interactions were identified. Eight patients (20.0%; 95% CI, 7.6% to 32.4%) had partial responses and 26 (65.0%; 95% CI, 50.2% to 79.8%) had stable disease as their best response. The median overall survival for the 34 patients treated at the phase II dose was 12.6 months, with progression-free survival of 6.2 months. These data compare favorably with conventional chemotherapy in the salvage setting for NCSLC where the response rates are < 10% and median survivals are 6-8 months (14-16).

In an attempt to improve the therapeutic index for initial therapy of metastatic NSCLC, the combination of bevacizumab and erlotinib is being proposed as first-line treatment in place of conventional chemotherapy. The regimen will be beneficial if toxicity is reduced and efficacy is unchanged or if efficacy is improved. Since this regimen causes no hair loss, minimal nausea and no cytopenia, which nearly eliminated the risks of infections and bleeding, the combination of targeted agents appears to be better tolerated than conventional chemotherapy. Efficacy may also be improved since its activity in the salvage setting when patients are less likely to respond to any treatment rivals that of conventional chemotherapy in the untreated setting. In addition, erlotinib alone in the untreated setting can yield results that are not dissimilar from chemotherapy under similar conditions. Hence, it is hypothesized that the combination of erlotinib plus bevacizumab can produce superior results with less toxicity. This trial is intended to provide pilot data for a future randomized trial of this combination of targeted agents versus conventional chemotherapy for advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria

* Histological or cytological diagnosis of non-squamous, non-small cell lung cancer. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible.
* Stage wet IIIB-IV or recurrent disease
* No significant hemoptysis (bright red blood< 1/2 teaspoon or more per episode within 3 months)
* Performance status of 0-1
* Prior radiation allowed if > 15 days.
* No prior treatment for metastatic disease. Adjuvant treatment allowed if greater than 6 months has passed.

Exclusion Criteria

Disease-Specific Exclusions

* History of hemoptysis (bright red blood of 1/2 teaspoon or more per episode) within 3 months prior to study enrollment.
* Current, ongoing treatment with full-dose warfarin
* Current or recent (within 10 days of enrollment) use of aspirin (>325 mg/day) or chronic use of other NSAIDs.
* Performance status =2-4
* Known HIV-related disease

General Medical Exclusions

Subjects meeting any of the following criteria are ineligible for study entry:

* Inability to comply with study and/or follow-up procedures
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study

Bevacizumab (Avastin®)-Specific Exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either
* Urine protein:creatinine (UPC) ratio > 1.0 at screening OR
* Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wallace Akerley, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Akerley W, Boucher K, Rich N, Egbert L, Harker G, Bylund J, Van Duren T, Reddy C. A phase II study of bevacizumab and erlotinib as initial treatment for metastatic non-squamous, non-small cell lung cancer with serum proteomic evaluation. Lung Cancer. 2013 Mar;79(3):307-11. doi: 10.1016/j.lungcan.2012.12.005. Epub 2012 Dec 25. PMID 23273522

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1:Bevacizumab and Erlotinib: Bevacizumab and Erlotinib: Erlotinib 150 mg/day orally plus bevacizumab 15 mg/kg intravenously every 21 days
Period: Overall Study
Arm/Group | Arm 1:Bevacizumab and Erlotinib
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Bevacizumab and Erlotinib: Erlotinib 150 mg/day orally plus bevacizumab 15 mg/kg intravenously every 21 days
Arm/Group | Arm 1
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Overall Survival
Description: The length of time from the start of treatment for a disease that patients are still alive.
Time Frame: 2 years
Population: All patients were included in response assessment based on intention to treat including those who received less than 6 weeks of therapy
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm 1:Bevacizumab and Erlotinib
Number analyzed (Participants) | 50
weeks | 50.4 [43.2 to 57.6]

2. Secondary Outcome: Evaluation of Progression-free Survival
Description: The length of time during and after bevacizumab-erlotinib that a patient lives with the disease but does not progress according to RECIST 1.0 Criteria. Per Response Evaluation Criteria In Solid Tumors (RECIST v1.0) for target lesions and assessed by CT: Progressive Disease (PD), >=20% increase in the sum of the longest diameter of target lesions
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm 1:Bevacizumab and Erlotinib
Number analyzed (Participants) | 50
weeks | 15.5 [13.3 to 17.7]

3. Secondary Outcome: Evaluation of Response Rate
Description: The percentage of patients in which response (CR + PR) was observed: Per Response Evaluation Criteria In Solid Tumors (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1:Bevacizumab and Erlotinib
Number analyzed (Participants) | 50
percentage of participants | 24 [12.2 to 35.8]

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 16/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=50)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
death (Investigations) | 2 (2)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture Bone-Hip (Musculoskeletal and connective tissue disorders) | 2 (2)
Hemmorrhage: Pulmonary (Blood and lymphatic system disorders) | 1 (1)
Infection: Abdomen (Infections and infestations) | 1 (1)
Infection: Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Lipase Elevated (Metabolism and nutrition disorders) | 1 (1)
Pain: Abdominal (Gastrointestinal disorders) | 1 (1)
Pain: Chest (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Reversibly Encephalopathy Syndrome (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=50)
Alkaline Phosphatase: Increased (Metabolism and nutrition disorders) | 10 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8)
ALT Increase (Metabolism and nutrition disorders) | 10 (16)
Anorexia (Gastrointestinal disorders) | 30 (38)
AST Increase (Metabolism and nutrition disorders) | 14 (17)
Ataxia (Nervous system disorders) | 4 (4)
Bruising (Skin and subcutaneous tissue disorders) | 3 (3)
Chills (Investigations) | 8 (8)
Confusion (Nervous system disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Creatinine Increased (Metabolism and nutrition disorders) | 7 (10)
Dehydration (Gastrointestinal disorders) | 11 (14)
Diarrhea (Gastrointestinal disorders) | 34 (56)
Dizziness (Nervous system disorders) | 6 (7)
Dry Mouth (Gastrointestinal disorders) | 4 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (19)
Edema (Blood and lymphatic system disorders) | 6 (6)
Fatigue (Investigations) | 24 (42)
Fever (Investigations) | 8 (10)
Anemia (Blood and lymphatic system disorders) | 6 (7)
Hemorrhage: Nose (Blood and lymphatic system disorders) | 9 (11)
Hemorrhage: Pulmonary (Blood and lymphatic system disorders) | 4 (4)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 7 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (13)
Hypertension (Cardiac disorders) | 6 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 11 (13)
Hypotension (Cardiac disorders) | 3 (3)
Infection: Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Infection: Urinary Tract (Renal and urinary disorders) | 6 (10)
Lymphopenia (Blood and lymphatic system disorders) | 9 (10)
Mood Alteration: Anxiety (Nervous system disorders) | 8 (8)
Mood Alteration: Depression (Nervous system disorders) | 5 (6)
Mucositis (Gastrointestinal disorders) | 12 (13)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 8 (8)
Nail Changes (Skin and subcutaneous tissue disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 21 (32)
Pain: Abdominal (Gastrointestinal disorders) | 7 (7)
Pain: Back (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain: Chest (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Pain: Headache (Nervous system disorders) | 4 (7)
Pain: Musculoskeletal Limb (Musculoskeletal and connective tissue disorders) | 14 (17)
Platelets: Decreased (Blood and lymphatic system disorders) | 7 (11)
Proteinuria (Metabolism and nutrition disorders) | 6 (11)
Rash (Skin and subcutaneous tissue disorders) | 43 (76)
Rash: Hand/Foot (Skin and subcutaneous tissue disorders) | 5 (5)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Serum Bicarbonate Decreased (Metabolism and nutrition disorders) | 5 (5)
Taste Alteration (dysgeusia) (Gastrointestinal disorders) | 9 (9)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 13 (20)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (15)
Weight Loss (Investigations) | 16 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes